CLINICAL TRIAL: NCT04448197
Title: The Real World Study on of Insomnia Treated by Traditional Chinese Medicine and Observation of Its Correlation With Circadian Rhythm
Brief Title: Insomnia Treated by Traditional Chinese Medicine and Its Circadian Rhythm
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Xiuqin Wang, Chief physician, The First Affiliated Hospital with Nanjing Medical University
Other Study IDs: 2019-SR-484
Record Dates: First submitted 2020-02-11; First posted 2020-06-25 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Traditional Chinese Medicine; Insomnia; Circadian Rhythm
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Routine blood test
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Chinese Medicine — Dialectical treatment of traditional Chinese medicine according to different constitution

SUMMARY:
Insomnia and sleep disorders are prominent health problems in modern society. High working pressure, fast pace of life, the use of electronic products and other reasons lead to the high incidence of insomnia and sleep disorders, which affect people's physical and mental health seriously, long-term insomnia will increase the risk of various health problems, and may even lead to malignant accidents. There are few effective methods to treat insomnia or sleep disorders, only part of the problem can be solved by sleeping pills and psychotherapy. However, drug therapy has side effects such as drowsiness on the next day, ataxia, anterograde amnesia and so on, and long-term application is addictive. Traditional Chinese medicine (TCM) has certain characteristics and advantages in the treatment of insomnia, but there is lack of evidence in clinical research that meets the requirements of modern evidence-based medicine, to prove the exact efficacy and safety of TCM in the treatment of insomnia. In addition, the research shows that the internal biological clock cycle of normal human body is 24-hour, insomnia may be related to biological clock gene. In this study, the outpatients with insomnia were taken as the research object. To observe the efficacy and safety of TCM in the treatment of insomnia by recording the participants' baseline demographic data, questionnaire survey, and conducting hematology examination. At the same time, to know the TCM constitution type of insomnia patients, through questionnaire survey with "Classification and Determination of TCM constitution table" that published by China Association of Chinese Medicine.And to explore the correlation between insomnia and circadian rhythm of biological clock .

DETAILED DESCRIPTION:
To record the demographic information and clinical characteristics of participants, including age, gender, education background, and drug use. Venous blood samples were collected and sent to laboratory test for blood routine, blood biochemistry, and blood homocysteine before and after 1 months of treatment. The remaining blood samples were kept in the sample bank for preservation. The Pittsburgh sleep quality index (PSQI) was used to evaluate the patients' sleep quality, and the depressive symptoms were assessed by Hamilton Depression Scale (HAMD-17) before and after treatment. Conduct the "Classification and Determination of TCM constitution table" before the treatment and 1-2 weeks before the end of the treatment, and according to the TCM constitution type to give constitution conditioning treatment.The participants will have a follow-up visit every two weeks, and the TCM will be adjusted according to the condition of illness. The treatment will last for 1 months.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients or inpatients.
* It conforms to the insomnia diagnosis standard of Chinese adult insomnia diagnosis and treatment guide (2017 Edition).
* Informed consent, voluntary participation in the study.

Exclusion Criteria:

* Sleep apnea syndrome leads to insomnia.
* Severe depression, suicidal tendency or having committed suicide.
* Pregnant and lactating women.
* It has serious primary heart, liver, lung, kidney, blood or serious diseases affecting its survival, such as: tumor or AIDS, SCR > 1.5n (n is the upper limit of normal value), ALT > 2n (n is the upper limit of normal value), WBC < 3.0 × 109 / L;
* Those who cannot give full informed consent due to mental disorders.
* According to the researcher's judgment, other situations that are not suitable for the group, such as the change of working environment and other vulnerable interviewers.
* Patients who are participating in other clinical studies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients or inpatients of The First Affiliated Hospital of Nanjing Medical University (Jiangsu Province Hospital) ，age 18-75 years old, male and female unlimited，in line with the Chinese adult insomnia diagnosis and treatment guidelines (2017 version) insomnia diagnosis standards， informed consent, voluntary participation in this study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the total score of the Pittsburgh sleep quality index (PSQI) at Month 1 | Baseline and month 1
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. Possible scores range from 0(the best sleep quality) to 21(the worst possible sleep quality).The higher the score of PSQI, the worse the sleep quality. Change=(Month 1 Score-Baseline Score)
Change from Baseline in the total score of the 17-item Hamilton Depression Scale (HAMD-17) at Month 1 | Baseline and month 1
  The 17-item Hamilton Depression Rating Scale(HAMD-17) assesses severity ranges of depression: no depression (0-7); mild depression (8-16); moderate depression (17-23); and severe depression (≥24). Possible scores range from 0(no depression) to 54(the worst possible depression). The higher the score of HAMD-17, the heavier the depression. Change=(Month 1 Score-Baseline Score)

SECONDARY OUTCOMES:
Change in of the ALT，to evaluate the safety of TCM treatment | Baseline and month 1
  Alanine aminotransferase, ALT in U/L.
Change in of the AST，to evaluate the safety of TCM treatment | Baseline and month 1
  Aspartate aminotransferase, AST in U/L
Change in of the BUN，to evaluate the safety of TCM treatment | Baseline and month 1
  Blood urea nitrogen, BUN in mmol/L
Change in of the Scr，to evaluate the safety of TCM treatment | Baseline and month 1
  Serum creatinine, Scr in μmol/L
Change in of the Hcy，to evaluate the safety of TCM treatment | Baseline and month 1
  Homocysteine, Hcy in μmol/L
Genome-wide association study，in bp，to explore the correlation between insomnia and circadian rhythm of biological clock | 1 year
  Illumina HumanHap550-Duo BeadChips was used to perform the whole genome genotyping in deCODE genetics (Reykjavı'k, Iceland)

CONTACTS AND LOCATIONS:
Overall Officials: Xiuqin Wang, doctor, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided